CLINICAL TRIAL: NCT06862622
Title: Task-based Synchronous Electroencephalography and Functional Magnetic Resonance Imaging (EEG-fMRI) to Explore Neural Representations of Memory Maintenance in the Aging Brain.
Brief Title: Neural Representations of Memory Transformation (MEM_TRANS)
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kirstin-Friederike Heise, Assistant Professor-Faculty, Medical University of South Carolina
Other Study IDs: Pro00141769
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Healthy Older Adults
Keywords: Aging; Healthy Volunteer Studies; memory; fMRI; EEG

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- behavioral skill learning intervention: All participants in this study undergo daily practice of a new skill until change through practice stabilizes (plateau).
  Interventions: Behavioral: Computer-based visuomotor sequence learning and interference

INTERVENTIONS:
Behavioral: Computer-based visuomotor sequence learning and interference — The behavioral sequence learning and interference paradigm allows the experimental manipulation of sequence memory after long-term consolidation achieved through individualized longitudinal practice and serves the extraction of the primary behavioral outcome. The learning task requires participants to respond with keypresses on a standard computer keyboard of visual targets. Participants will implicitly (without being made aware) learn sequential regularities provided through the recurring order of cued keys contrasted with random keys. Participants will practice the learning task remotely over consecutive days until a stable performance plateau is reached. During this phase, data will be collected online, and behavioral change will be monitored in real time. Then participants will undergo the behavioral interference intervention, in which the initially learned sequence memory will be perturbed through (implicit) exposure to new sequential information (i.e., interference).

SUMMARY:
Investigators overarching goal is to provide evidence for the link between altered spatiotemporal (where and when) neural mechanisms and the extent of changed memory maintenance in healthy older adults and to identify potential neural markers of compensatory function (cognitive resource). Investigators preliminary studies suggest that healthy older adults, compared to younger adults, benefit behaviorally from increased coupling between frontal and parietal brain waves when retrieving and updating well-consolidated visuomotor sequence memory via stronger top-down cognitive control of memory maintenance. Thus, Investigators central hypothesis is that the dynamics across cortical and subcortical regions (i.e., spatiotemporal representations) during transitions between different levels of memory stability indicate the efficiency of memory maintenance. The rationale is that while temporal and spatial neural signatures carry distinct mechanistic information, the joint definition of spatial and temporal representations will allow the differentiation of compensatory versus neurodegenerative mechanisms.

DETAILED DESCRIPTION:
To investigate the spatiotemporal neural dynamics during memory maintenance mechanisms, healthy older adults will practice a computer-based online visuomotor sequence learning task over consecutive days until reaching a performance plateau. At the performance plateau, participants will undergo concurrent electroencephalography and magnetic resonance imaging (EEG-fMRI) while being exposed to a behavioral interference intervention to perturb the stability of the previously stored memory trace to extract spatiotemporal neural dynamics during these transitional states. Additionally, participants will undergo an additional brain scan to quantify aging-related neurodegeneration based on grey- and white-matter integrity, cerebral perfusion, and resting-state connectivity. Cognitive functioning and putative confounders of learning and memory will be quantified with standardized assessments. The experimental procedures include an individual number of daily computer-based sessions of task practice at home, and two lab visits including questionnaires, neuropsychological testing, and two MRI brain scans distributed over approximately two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older (80 of the final sample will be ≥60years of age)
* Cognitively unimpaired, ambiguous, or mildly impaired cognitive function, defined as a score of ≥18 in the Montreal Cognitive Assessment (MOCA).
* No previous stroke, brain tumor, neurodegenerative disease, or trauma to the head
* Ability to give consent for study participation
* Ability to perform a computer task requiring responding to visual cues and typing on a standard computer keyboard with both index and middle fingers for 30 minutes daily.

Exclusion Criteria:

* Inability to use both index and middle fingers to type on a standard computer keyboard
* Dementia defined as a score of <18 in the Montreal Cognitive Assessment (MOCA)
* Uncorrected vision, hindering perception of visual cues presented on a standard computer screen
* Medication use at the time of study that may interfere with learning, including but not limited to carbamazepine, flunarizine, sulpiride, rivastigmine, and dextromethorphan.
* Neuromuscular disorders that affect fine motor control of the hands.
* Presence of neurological or psychiatric disorders
* Presence of scalp injury or disease
* Prior intracranial surgery
* Prior brain radiotherapy
* Prior history of intracranial tumor, intracranial infection, or cerebrovascular malformation
* Metal in the head or neck
* Contraindications to MRI (such as severe claustrophobia, implanted medical devices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers aged18 years or older (80 of the final sample will be ≥60years of age).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in relative performance precision | 60 minutes
  The primary behavioral outcome parameter is based on the precision of keypresses, i.e., temporal and spatial deviation of pressed from cued keys measured in a single compound measure [actual precision in %] serve to describe behavior across retrieval of formerly consolidated and interference with competing new sequential information.
Whole-brain change in time-resolved neural dynamics extracted EEG (temporal representations). | 60 minutes
  Temporal patterns of brain dynamics derived from electroencephalography and projected into the anatomical source space serve to describe the temporal representations across retrieval of formerly consolidated and interference with competing new sequential information.
Change in blood-oxygenation-level-dependent (BOLD) derived brain activation patterns (spatial representations) | 60 minutes
  Change of spatially precise whole-brain blood-oxygenation-level-dependent (BOLD) signal changes (spatial representations) across retrieval of formerly consolidated and interference with competing new sequential information.

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin-Friederike Heise, PhD, Principal Investigator — Medical University of South Carolina